CLINICAL TRIAL: NCT00939042
Title: Percutaneous Intramyocardial Cell Therapy After Acute Myocardial Infarction Using Bone Marrow Mononuclear Cells
Brief Title: Alster Stem Cells - Intramyocardial Stem Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: Asklepios proresearch (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1777; 2008-004625-42 (EudraCT Number)
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Acute Myocardial Infarction; Early Left Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): PCI plus BNNC Therapy after acute myocardial infarction
  Interventions: Procedure: BMNC therapy
- 2 (Active Comparator): Percutaneous Coronary Intervention after acute myocardial infarction
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — common Percutaneous Coronary Intervention
  Arms: 2
Procedure: BMNC therapy — Injection of BMNC after common PCI
  Arms: 1

SUMMARY:
Study to assess the efficacy of intramyocardial bone marrow derived mononuclear cell therapy concerning left ventricular ejection fraction as measured by echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* LVDF < 45% after timely (max. 6 hours after the onset of symptomps) successful PCI
* conventional therapy according to the ESC guidelines for heart failure
* BMI > 20 and < 35

Exclusion Criteria:

* PCI elder then 21 days
* relevant valvular disease
* history of stroke/multivessel disease/thromboembolic event etc.
* DM Type I
* pregancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the effect of a direct intramyocardial injection of bone marrow mononuclear cells (BMNC) on heart function (LVEF). | 12 months

SECONDARY OUTCOMES:
Comparison of th eexplanatory power of echocardiography, endocardial left ventricular electromechanical mapping (LVEMM) with NOGA and cardiac MRI as an endpoint for myocardial regeneration. | 12 months
Collection of first evidence on the best type and time points for the determination of myocardial regeneration by NOGA and other parameters. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Kuck, MD, PhD, Principal Investigator — Asklepios Klinik St. Georg, Department of Cardiology
Locations (1):
- Asklepios Klinik St. Georg, Hamburg, Germany